CLINICAL TRIAL: NCT04790630
Title: Cognitive Remediation of Cognitive Control in Late-Life Depression
Brief Title: Cognitive Fitness for Depression in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kevin Manning, Associate Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-046-2; 1K23MH118420-01A1 (NIH)
Record Dates: First submitted 2021-01-13; First posted 2021-03-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-04

CONDITIONS: Depression Mild; Depressive Disorder, Major; Mild Cognitive Impairment
MeSH Terms: conditions — Depressive Disorder, Major; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computerized Cognitive Remediation of Executive Functioning (CCR-EF) (Experimental): Initially 10 hours of processing speed exercises from "Brain HQ", (the 3 exercises are auditory tone sweep, visual processing [Double Decision], visual sweep).
  Following the 8-10 hours of Brain HQ, participants complete 8-10 hours of "Ultimate Word Master" before completing 16-20 hours of "Neurogrow" (formerly called "Catch the Ball").
  Participants are asked to complete approximately 28-42 hours of computerized brain training over 4-6 weeks.
  Interventions: Other: Computerized Cognitive Remediation of Executive Functioning (CCR-EF)
- Active Control (Active Comparator): Patients in the active control arm will complete three activities according to a standard protocol: 1) play a visuospatially oriented computer game (Myst), 2) watch computer-based educational programs on art, history, literature, and 3) play computer games online through the Brain HQ platform; games include crossword puzzles, soduko, paddleboard, and word search. Participants will complete a total of 32-42 hours of training over 4-6 weeks. Time spent on each task will be evenly divided (15 minutes of each task everday).
  Interventions: Other: Active Control

INTERVENTIONS:
Other: Computerized Cognitive Remediation of Executive Functioning (CCR-EF) — computerized experimental brain-training treatment
  Arms: Computerized Cognitive Remediation of Executive Functioning (CCR-EF)
Other: Active Control — computerized intervention that follows recommendations for cognitive fitness
  Arms: Active Control

SUMMARY:
This research is being done to determine if computerized administered cognitive fitness activities will improve thinking and depression in older depressed adults who are being treated with antidepressants. The investigators are also interested in whether participating in the treatment will result in changes to brain activity measured with magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
Major depression in the elderly is both challenging to treat and detrimental to the cognitive functioning of patients. Major depression increases the probability of a later dementia diagnosis. By targeting cognitive processes in treatment, the investigators hope to both find a more effective means to manage major depression in older adults, but also demonstrate how top-down processes (e.g., Executive Control Network) may be driving depression and cognitive decline in older adults.

The investigators are recruiting older adults with and without mild cognitive impairment. All subjects must have at least mild depressive symptoms to be eligible to participate. Subjects will be randomly assigned to one of two different interventions.

Results of this study will help the investigators understand the mechanisms that contribute to depressed mood and cognitive change in older adults with late life depression.

ELIGIBILITY:
Inclusion Criteria:

* ability to read and write in English
* current major or mild depression despite ongoing treatment
* under the care of a physician who prescribes medication for depression
* currently treated with an antidepressant for at least 8 weeks

Exclusion Criteria:

* psychosis
* other psychiatric disorders (except personality & generalized anxiety disorders)
* substance use disorders in the prior year
* clinical diagnosis of dementia
* neurological disorders (e.g., stroke, epilepsy, brain injury with loss of consciousness > 30 minutes, brain tumors, demyelinating diseases)
* corrected visual acuity < 20/70 or color blindness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Change in attention / cognitive flexibility as measured by the Trail Making Part B test | Pre-treatment and six weeks later when treatment has ended
  time to complete alpha-numeric sequencing
Change in depression symptom severity as measured with the Montgomery Asberg Depression Rating Scale (MADRS) | Pre-treatment and six weeks later when treatment has ended
  depression rating scale

SECONDARY OUTCOMES:
Change in verbal learning as measured with the California Verbal Learning Test (CVLT) Total Learning | Pre-treatment and six weeks later when treatment has ended
  number of words recalled over 5 trials and spontaneous semantic organization of those words
Change in attention processing speed as measured with the Flanker Test of Response Inhibition from the NIH Cognitive Toolbox | Pre-treatment and six weeks later when treatment has ended
  computerized test of response inhibition, speed of responding
Change in self-reported depressive symptoms measured with the Carroll Depression Rating Scale | Pre-treatment and six weeks later when treatment has ended
  self-report of depression symptoms
Change in problem solving/speed/spatial memory as measured with the NIH Toolbox fluid composite scales | Pre-treatment and six weeks later when treatment has ended
  computerized picture memory, simple processing speed, problem solving/mental flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Manning, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP, ICF
Time Frame: Data will be available March 2025